CLINICAL TRIAL: NCT00528892
Title: An Open-label, Randomized, 48-Week Study to Assess the Safety, Tolerability and Activity of Raltegravir When Replacing the Ritonavir-boosted PI Component of HAART in HIV-Infected Individuals With Viral Load Suppression on a Ritonavir-Boosted PI Containing Regimen.
Brief Title: Switching From PI to RALtegravir in HIV Stable Patients
Acronym: SPIRAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Jose M Gatell, Hospital Clinic barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPIRAL; EUDRACT: 2007-003401-27
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2008-05

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Switch current boosted-PI to raltegravir 400 mg BID.
  Interventions: Drug: Raltegravir
- 2 (Active Comparator): Continue current regimen (ritonavir-boosted PI plus at least 2 other drugs)
  Interventions: Drug: boosted PI

INTERVENTIONS:
Drug: Raltegravir — switching PI to raltegravir
  Arms: 1
Drug: boosted PI — continue on boosted-PI
  Arms: 2

SUMMARY:
The investigators hypothesis is that switching from a ritonavir-boosted PI to raltegravir may be associated with an at least non-inferior effectiveness, virological response and safety, and even a better tolerability profile with regard to lipid metabolism, insulin resistance, body fat distribution as compared with continuation of the baseline regimen in HIV-1 seropositive males or females at least 18 years of age and older on ritonavir-boosted PI plus at least 2 other drugs and plasma viral RNA below 50 copies/mL.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a male or female at least 18 years of age.
* Women of childbearing potential must have a negative serum pregnancy test (HCG) within 10 days prior to randomization into the study.
* Patients must use adequate birth control measures (barrier method.)
* Patients must be HIV 1 seropositive using standard diagnostic criteria.
* Patients must have two plasma viral RNA measurements below detection limits with the routine ultrasensitive method used at each participating site (at least <50 copies/mL) within 180 days prior to randomization into this study.
* Patients must be on continuous therapy with HAART consisting of a ritonavir-boosted protease-inhibitor (PI) and at least two other antiretroviral agents for at least 6 months prior to randomization into this study, with no planned drug changes in the following 12 months. Boosted PIs can be indinavir, fosamprenavir, saquinavir, lopinavir, atazanavir, tipranavir or darunavir.
* Patients must be considered clinically stable, in the opinion of the investigator, at the time of entry into the study; i.e., clinical status and all chronic medications should be unchanged for at least 14 days prior to randomization. Patients currently receiving treatment for an opportunistic infection may be allowed into the study as long as the above criteria are met. Prophylaxis for opportunistic infections consistent with standard treatment is permissible. .
* The following laboratory values must be obtained within 2-4 weeks of randomization into the study:

  * Hemoglobin >8.0 g/dL.
  * Absolute neutrophil count > 750/mm3
  * Platelet count > 50,000/ mm3
  * Creatinine < 2.0 mg/dL.
  * Transaminases (ALAT, ASAT) <5xULN

Exclusion Criteria:

* Pregnancy or breast feeding or women planning pregnancy during the study duration.
* Patients on ART regimens not likely to be maintained during the whole study duration
* Prior use of HIV integrase inhibitors.
* Use of any investigational agents (other than ART on expanded access programme) within 90 days of randomization.
* Alcohol or substance abuse which in the opinion of the investigator would interfere with patient compliance or safety.
* Patients with an active opportunistic infection or malignancy. Patients with a chronic, stable opportunistic infection will be allowed to enter this study.
* Any condition or history of any illness which, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering the study drugs to the patient.
* Any patient with a diagnosis of visceral Kaposi's sarcoma. Patients with lymphedema secondary to cutaneous Kaposi's sarcoma, or with cutaneous or palatal Kaposi's sarcoma that has been treated with systemic immunosuppressive therapy must also be excluded.
* Any patient with a diagnosis of acute hepatitis due to any cause. Patients with chronic hepatitis including chronic hepatitis B surface antigenemia chronic hepatitis C may enter the study as long as they have stable liver function tests and meet all inclusion criteria. Patients with acute exacerbations of chronic hepatitis are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with treatment failure (i.e.: those with viral failure, developing new CDC-C events, switching assigned treatment for any cause, withdrawing consent, being lost to follow-up or dying) | 48 weeks

SECONDARY OUTCOMES:
The proportion of patients with viral failure while on assigned treatment (defined as two consecutive plasma HIV-RNA below detection limits) | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Gatell, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Saumoy M, Sanchez-Quesada JL, Martinez E, Llibre JM, Ribera E, Knobel H, Gatell JM, Clotet B, Curran A, Curto J, Maso M, Ordonez-Llanos J, Podzamczer D. LDL subclasses and lipoprotein-phospholipase A2 activity in suppressed HIV-infected patients switching to raltegravir: Spiral substudy. Atherosclerosis. 2012 Nov;225(1):200-7. doi: 10.1016/j.atherosclerosis.2012.08.010. Epub 2012 Sep 6. PMID 23017355
- [Derived] Martinez E, Larrousse M, Llibre JM, Gutierrez F, Saumoy M, Antela A, Knobel H, Murillas J, Berenguer J, Pich J, Perez I, Gatell JM; SPIRAL Study Group. Substitution of raltegravir for ritonavir-boosted protease inhibitors in HIV-infected patients: the SPIRAL study. AIDS. 2010 Jul 17;24(11):1697-707. doi: 10.1097/QAD.0b013e32833a608a. PMID 20467288